CLINICAL TRIAL: NCT01573559
Title: ClearView Predicate Comparison Testing
Status: Completed | Type: Observational
Sponsor: Epic Research & Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EPIC-003
Record Dates: First submitted 2011-10-03; First posted 2012-04-09 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Ambulatory adults with no apparent health conditions

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ClearView/Predicate

SUMMARY:
This study serves as a comparison study between the EPIC ClearView and a predicate device.

DETAILED DESCRIPTION:
The EPIC ClearView is a galvanic skin response (GSR) measurement system that is intended to be used to determine autonomic response as psychological indicators by measuring the electrical resistance of the skin. The EPIC ClearView is a non-invasive digital bioelectrography instrument that is used to assess the electrophysiology of humans. The measurements are digital photographs taken in a brief exposure to an electric field. These measurements are quantified to produce a standardized Response Scale.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male or Female.
* Age range: 18 to 85.
* The subject is able to understand and provide signed consent for the procedure.
* Every effort will be given to balance subjects by gender, age, and race.

Exclusion Criteria:

* Subjects < 18 years in age or > 85 years in age.
* Inability or unwillingness to provide informed consent.
* Subjects with pacemakers or another electrical device, such as an automatic internal cardiac defibrillator, implanted somewhere in their body.
* Subjects missing all or part of any of their fingers.
* Subjects with hand tremors or involuntary oscillations ("shaking") of the hands that prevent clear imaging.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women ages 18-85.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Correlation Between ClearView and Predicate | At time of study scan (Single study visit only, with no follow-up. The study endpoint will be reported for day 0, the day of the study visit.)
  The primary objective of this study is to perform a point-to-point comparison of the EPIC ClearView™ galvanic skin response hand measurements (on a 0-25 scale) to those of a predicate device (on a 0-100 scale). We hypothesize that there will be a statistically significant correlation between the galvanic skin response measurements made by the two devices.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Rizzo, PhD, Principal Investigator — Epic Research & Diagnostics, Inc.
Locations (1):
- EPIC Research & Diagnostics, Inc., Scottsdale, Arizona, United States